CLINICAL TRIAL: NCT05629585
Title: A Phase 3 Open-label, Randomised Study of Datopotamab Deruxtecan (DatoDXd) With or Without Durvalumab Versus Investigator's Choice of Therapy in Patients With Stage I-III Triple-negative Breast Cancer Who Have Residual Invasive Disease in the Breast and/or Axillary Lymph Nodes at Surgical Resection Following Neoadjuvant Systemic Therapy (TROPION-Breast03)
Brief Title: A Study of Dato-DXd With or Without Durvalumab Versus Investigator's Choice of Therapy in Patients With Stage I-III Triple-negative Breast Cancer Without Pathological Complete Response Following Neoadjuvant Therapy (TROPION-Breast03)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo (Industry); SWOG Clinical Trials Partnerships (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D926XC00001; 2023-505552-22-00 (Registry Identifier: CTIS (EU)); 2022-002680-30 (EudraCT Number)
Record Dates: First submitted 2022-11-04; First posted 2022-11-29 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; TNBC; Triple-negative; Adjuvant; Datopotamab Deruxtecan; Dato-DXd; DS1062a; Antibody Drug Conjugate; ADC; TROP2; Durvalumab
MeSH Terms: conditions — Breast Neoplasms | interventions — durvalumab; Capecitabine; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Parallel
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dato-DXd in combination with Durvalumab (Experimental): Arm 1: Dato-DXd 6 mg/kg IV Q3W x 8 cycles + Durvalumab 1120 mg IV Q3W x 9 cycles
  Interventions: Drug: Dato-DXd; Drug: Durvalumab
- Dato-DXd (Experimental): Arm 2: Dato-DXd 6 mg/kg IV Q3W x 8 cycles
  Interventions: Drug: Dato-DXd
- Investigators Choice Therapy (Active Comparator): Arm 3: Capecitabine (1000 or 1250 mg/m2 oral BID on Days 1 to 14, Q3W) for 8 cycles
  Pembrolizumab* (200 mg IV on Day 1, Q3W) for 9 cycles
  Capecitabine (1000 or 1250 mg/m2 oral BID on Days 1 to 14, Q3W) for 8 cycles + pembrolizumab* (200 mg IV on Day 1, Q3W) for 9 cycles
  * Only participants who have received prior pembrolizumab in the neoadjuvant setting should receive pembrolizumab as part of their adjuvant therapy on Arm 3.
  Interventions: Drug: Capecitabine; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Dato-DXd — Experimental drug. Provided in 100mg vials. IV infusion
  Other Names: Datopotamab deruxtecan (Dato-DXd, DS-1062a)
  Arms: Dato-DXd; Dato-DXd in combination with Durvalumab
Drug: Durvalumab — Experimental drug. Provided in 50mg vials. IV infusion
  Other Names: MEDI4736
  Arms: Dato-DXd in combination with Durvalumab
Drug: Capecitabine — Active Comparator. Tablet. Oral route of administration
  Other Names: XELODA®, Capecitabine Cell Pharm, Capecitabine EG, Capecitabine Accord
  Arms: Investigators Choice Therapy
Drug: Pembrolizumab — Active Comparator. Provided in 100mg vials. IV infusion
  Other Names: KEYTRUDA®
  Arms: Investigators Choice Therapy

SUMMARY:
This is a Phase III, randomized, open-label, 3-arm, multicenter, international study assessing the efficacy and safety of Dato-DXd with or without durvalumab compared with ICT in participants with stage I to III TNBC with residual invasive disease in the breast and/or axillary lymph nodes at surgical resection following neoadjuvant systemic therapy.

DETAILED DESCRIPTION:
The study will investigate the efficacy and safety of Dato-DXd with or without durvalumab when compared with ICT (capecitabine and/or pembrolizumab) in participants with stage I to III TNBC who have residual invasive disease in the breast and/or axillary lymph nodes at surgical resection following neoadjuvant systemic therapy.

The primary objective of the study is to demonstrate superiority of Dato-DXd in combination with durvalumab relative to ICT by assessment of iDFS in participants with stage I to III TNBC with residual invasive disease at surgical resection following neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥ 18 years at the time of screening.
2. Histologically confirmed invasive TNBC, as defined by the ASCO/CAP guidelines.
3. Residual invasive disease in the breast and/or axillary lymph node(s) at surgical resection following neoadjuvant therapy.
4. Completed at least 6 cycles of neoadjuvant therapy containing an anthracycline and/or a taxane with or without platinum chemotherapy, with or without pembrolizumab.
5. No evidence of locoregional or distant relapse.
6. Surgical removal of all clinically evident disease in the breast and lymph nodes.
7. ECOG performance status of 0 or 1 with no deterioration over the previous 2 weeks prior to randomisation.
8. All participants must provide an FFPE tumour sample from residual invasive disease at surgery for tissue-based analysis.
9. No adjuvant systemic therapy.
10. Radiotherapy (if indicated) delivered before the start of study intervention.
11. If post-operative radiation therapy is given, an interval of no more than 6 weeks between the completion of radiation therapy and the date of randomisation (radiation therapy can be completed during screening period). If no post-operative radiation therapy is given, an interval of no more than 16 weeks between the date of breast surgery and the date of randomisation.
12. Has LVEF ≥ 50% by either an ECHO or MUGA scan within 28 days before randomisation.
13. Eligible for one of the therapy options listed as investigator's choice per investigator assessment.
14. No known germline BRCA1 or BRCA2 pathogenic mutation.
15. Adequate bone marrow reserve and organ function within 7 days before randomisation.

Exclusion Criteria:

1. Stage IV (metastatic) TNBC.
2. History of prior invasive breast cancer, or evidence of recurrent disease following preoperative therapy and surgery.
3. Severe or uncontrolled medical conditions including systemic diseases, history of allogeneic organ transplant and active bleeding diseases, ongoing or active infection, serious chronic gastrointestinal conditions associated with diarrhea chronic diverticulitis or previous complicated diverticulitis.
4. History of another primary malignancy except for adequately resected basal cell carcinoma of the skin or squamous cell carcinoma of the skin, in situ disease (including ductal carcinoma in situ) that has undergone potentially curative therapy, or other solid malignancy treated with curative intent with no known active disease within 5 years before randomisation and of low potential risk for recurrence.
5. Persistent toxicities caused by previous anticancer therapy, excluding alopecia, not yet improved to Grade ≤ 1 or baseline. Participants with irreversible toxicity that is not reasonably expected to be exacerbated by study intervention may be included (eg, hearing loss).
6. Active or prior documented autoimmune or inflammatory disorders.
7. Clinically significant corneal disease.
8. Active or uncontrolled hepatitis B or C virus infection.
9. Known HIV infection that is not well controlled
10. Active tuberculosis infection.
11. Mean resting corrected QTcF > 470 ms regardless of gender, obtained from triplicate 12-lead ECGs performed at screening.
12. Uncontrolled or significant cardiac disease.
13. History of non-infectious ILD/pneumonitis including radiation, pneumonitis that required steroids, has current ILD/pneumonitis, or has suspected ILD/pneumonitis that cannot be ruled out by imaging at screening.
14. Has severe pulmonary function compromise.
15. Any known active liver disease.
16. Grade ≥ 2 peripheral neuropathy of any aetiology.
17. Prior exposure to a PD-1/PD-L1 inhibitor other than pembrolizumab.
18. Current or prior use of immunosuppressive medication within 14 days prior to randomisation.
19. Participants with a known severe hypersensitivity to Dato-DXd or any of the excipients of these products including but not limited to polysorbate 80 or other monoclonal antibodies.
20. Participants with a known severe hypersensitivity to PD-1/PD-L1 inhibitors.
21. Participation in another clinical study with a study intervention or investigational medicinal device administered in the last 4 weeks prior to randomisation, randomisation into a prior Dato-DXd, T-DXd, or durvalumab study regardless of treatment assignment.
22. Currently pregnant (confirmed with positive pregnancy test), breastfeeding or planning to become pregnant.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1174 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2027-09-20 (Estimated); Study Completion 2030-01-30 (Estimated)

PRIMARY OUTCOMES:
Invasive disease-free survival (iDFS) for Dato-DXd + durvalumab vs. ICT | From randomisation to date of the event, up to 57 months from first subject in
  iDFS is defined as time from randomisation until date of first occurrence of one of the following events: ipsilateral invasive breast tumour (local) recurrence, regional invasive breast cancer recurrence (axilla, regional lymph nodes, chest wall, and skin of ipsilateral breast), or distant recurrence (metastatic breast cancer that has either been biopsy-confirmed or clinically diagnosed as recurrent invasive breast cancer); contralateral invasive breast cancer; second primary non-breast invasive cancer (other than squamous or basal cell skin cancer); or death from any cause.
  iDFS will be determined based on disease recurrence per investigator assessment based on all available clinical assessments. The analysis will include all randomised participants, as randomised, regardless of whether the participant withdraws from randomised therapy or receives another anticancer therapy.
  The measure of interest will be the HR (hazard ratio) of iDFS for Dato-DXd + durvalumab vs ICT.

SECONDARY OUTCOMES:
Distant disease-free survival (DDFS) for Dato-DXd + durvalumab vs ICT | From randomisation to date of the event, up to 57 months from first subject in
  DDFS is defined as time from randomisation to date of first distant recurrence, occurrence of second primary non-breast invasive cancer, or death from any cause.
  DDFS is determined based on disease recurrence per investigators assessment based on all available clinical assessments.
  The analysis will include all randomised participants, as randomised regardless of whether the participant withdraws from randomised therapy or received another anticancer therapy. The measure of interest will be the HR (hazard ratio) of DDFS for Dato-DXd + durvalumab vs ICT.
DDFS for Dato-DXd vs ICT | From randomisation to date of the event, up to 57 months from first subject in
  DDFS is defined as time from randomisation to date of first distant recurrence, occurrence of second primary non-breast invasive cancer, or death from any cause. DDFS is determined based on disease recurrence per investigators assessment based on all available clinical assessments. The measure of interest will be the HR (hazard ratio) of DDFS for Dato-DXd vs ICT.
DDFS for Dato-DXd + durvalumab vs Dato-DXd | From randomisation to date of the event, up 57 months from first subject in
  DDFS is defined as time from randomisation to date of first distant recurrence, occurrence of second primary non-breast invasive cancer, or death from any cause. DDFS is determined based on disease recurrence per investigators assessment based on all available clinical assessments. The measure of interest will be the HR (hazard ratio) of DDFS for Dato-DXd + durvalumab vs Dato-DXd.
Overall Survival (OS) for Dato-DXd + durvalumab vs ICT | From randomisation to date of death, due to any cause, up to 87 months from first subject in
  OS is defined as time from randomisation until date of death due to any cause.
  The analysis will include all randomised participants, as randomised regardless of whether the participant withdraws from randomised therapy or received another anticancer therapy. The measure of interest will be the HR (hazard ratio) of OS for Dato-DXd + durvalumab vs ICT.
OS for Dato-DXd vs ICT | From randomisation to date of death, due to any cause, up to 87 months from first subject in
  OS is defined as time from randomisation until date of death due to any cause. The measure of interest will be the HR (hazard ratio) of OS for Dato-DXd vs ICT.
iDFS for Dato-DXd vs ICT | From randomisation to date of the event, up to 57 months from first subject in
  iDFS is defined as time from randomisation until date of first occurrence of one of the following events: ipsilateral invasive breast tumour (local) recurrence, regional invasive breast cancer recurrence (axilla, regional lymph nodes, chest wall, and skin of ipsilateral breast), or distant recurrence (metastatic breast cancer that has either been biopsy-confirmed or clinically diagnosed as recurrent invasive breast cancer); contralateral invasive breast cancer; second primary non-breast invasive cancer (other than squamous or basal cell skin cancer); or death from any cause.
  iDFS will be determined based on disease recurrence per investigator assessment based on all available clinical assessments. The analysis will include all randomised participants, as randomised, regardless of whether the participant withdraws from randomised therapy or receives another anticancer therapy.
  The measure of interest will be the HR (hazard ratio) of iDFS for Dato-DXd vs ICT.
iDFS for Dato-DXd + durvalumab vs Dato-DXd | From randomisation to date of the event, up to 57 months from first subject in
  iDFS is defined as time from randomisation until date of first occurrence of one of the following events: ipsilateral invasive breast tumour (local) recurrence, regional invasive breast cancer recurrence (axilla, regional lymph nodes, chest wall, and skin of ipsilateral breast), or distant recurrence (metastatic breast cancer that has either been biopsy-confirmed or clinically diagnosed as recurrent invasive breast cancer); contralateral invasive breast cancer; second primary non-breast invasive cancer (other than squamous or basal cell skin cancer); or death from any cause. The measure of interest will be the HR (hazard ratio) of iDFS for Dato-DXd + durvalumab vs Dato-DXd.
Participant-reported physical function in participants treated with Dato-DXd with or without durvalumab compared with ICT | From randomisation to date of the deterioration, up to 36 months after randomisation
  Time to Deterioration (TTD) and actual scores in physical function as measured by the PROMIS Physical Function Short Form 8c.TTD is defined as time from the date of randomisation to the date of deterioration. Deterioration is defined as change from baseline that reaches a clinically meaningful deterioration threshold.
  The analysis will include all dosed participants. The measure of interest is the HR (hazard ratio) of TTD and mean between-arm difference in physical function for Dato-DXd with or without durvalumab compared with ICT.
Participant-reported in GHS/QoL in participants treated with Dato-DXd with or without durvalumab compared with ICT | From randomisation to date of the deterioration, up to 36 months after randomisation
  Time to Deterioration (TTD) and actual scores in GHS/QoL as measured by the GHS/QoL scale from the EORTC IL172.
  TTD is defined as time from the date of randomisation to the date of deterioration. Deterioration is defined as change from baseline that reaches a clinically meaningful deterioration threshold.
  The analysis will include all randomised participants. The measure of interest is the HR (hazard ratio) of TTD and mean between-arm difference in GHS/QoL for Dato-DXd with or without durvalumab compared with ICT.
Participant-reported fatigue in participants treated with Dato-DXd with or without durvalumab compared with ICT | From randomisation to 24 months after randomisation
  Proportion of participants experiencing different levels of fatigue at 3 months (13weeks), 6 months (26 weeks), and 12 months (52 weeks) as measured by PROMIS Fatigue Short Form 7a.
  The analysis will include all dosed participants. The measure of interest will be the proportion of participants reporting different levels of fatigue.
Pharmacokinetics of Dato-DXd | Day 1 of cycles 1,2,4,6,8 (Each cycle is 21 days)
  Concentration of Dato- DXd, total anti-TROP2 antibody, and MAAA-1181 in plasma.
Immunogenicity of Dato-DXd | Day 1 of cycles 1,2,4,6,8 (Each cycle is 21 days) and within 35 days of completion of or discontinuation of study intervention (at an average of 6 months following randomization)
  Presence of ADAs for Dato-DXd (confirmatory results: positive or negative; titres).
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | Randomization to final safety follow-up visit, either 90 days after last dose of study intervention for those who complete planned study intervention or 90 days after date of discontinuation for those who discontinue study intervention prematurely
  Safety and tolerability will be evaluated in terms of AEs (graded by CTCAE version 5.0).

CONTACTS AND LOCATIONS:
Locations (228):
- United States (72):
  - Research Site, Gilbert, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Hot Springs, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Springdale, Arkansas
  - Research Site, Beverly Hills, California
  - Research Site, Costa Mesa, California
  - Research Site, Duarte, California
  - Research Site, Fountain Valley, California
  - Research Site, Irvine, California
  - Research Site, La Jolla, California
  - Research Site, Lakewood, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, Orange, California
  - Research Site, Roseville, California
  - Research Site, Upland, California
  - Research Site, Vallejo, California
  - Research Site, Denver, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Altamonte Springs, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Athens, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Maywood, Illinois
  - Research Site, Westwood, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Annapolis, Maryland
  - Research Site, Baltimore, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Camden, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Hershey, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Germantown, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Bedford, Texas
  - Research Site, Dallas, Texas
  - Research Site, Denton, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, McAllen, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Gainesville, Virginia
  - Research Site, Midlothian, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Edmonds, Washington
  - Research Site, Issaquah, Washington
  - Research Site, Puyallup, Washington
  - Research Site, Seattle, Washington
  - Research Site, Spokane Valley, Washington
  - Research Site, Morgantown, West Virginia
- Belgium (10):
  - Research Site, Anderlecht
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Hasselt
  - Research Site, Liège
  - Research Site, Namur
  - Research Site, Sint-Niklaas
  - Research Site, Wilrijk
- Brazil (6):
  - Research Site, Brasília
  - Research Site, Porto Alegre
  - Research Site, Recife
  - Research Site, Salvador
  - Research Site, São Paulo
  - Research Site, Vitória
- Canada (10):
  - Research Site, North Vancouver, British Columbia
  - Research Site, Barrie, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saskatoon, Saskatchewan
- China (25):
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenzhen
  - Research Site, Shijiazhuang
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xiamen
  - Research Site, Zhengzhou
- Denmark (6):
  - Research Site, Copenhagen
  - Research Site, Herning
  - Research Site, Næstved
  - Research Site, Odense
  - Research Site, Sønderborg
  - Research Site, Vejle
- France (11):
  - Research Site, Angers
  - Research Site, Bordeaux
  - Research Site, Dijon
  - Research Site, Lyon
  - Research Site, Montpellier
  - Research Site, Nîmes
  - Research Site, Paris
  - Research Site, Poitiers
  - Research Site, Rennes
  - Research Site, Saint-Herblain
  - Research Site, Villejuif
- Germany (16):
  - Research Site, Frankfurt am Main
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heilbronn
  - Research Site, Kiel
  - Research Site, Langen
  - Research Site, Leipzig
  - Research Site, Ludwigsburg
  - Research Site, Mönchengladbach
  - Research Site, München
  - Research Site, Paderborn
  - Research Site, Regensburg
  - Research Site, Stuttgart
  - Research Site, Troisdorf
  - Research Site, Tübingen
  - Research Site, Wuppertal
- Greece (3):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Thessaloniki
- Italy (12):
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Livorno
  - Research Site, Meldola
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Roma
  - Research Site, Rozzano
- Japan (23):
  - Research Site, Akashi-shi
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Hiroshima
  - Research Site, Isehara-shi
  - Research Site, Kashiwa
  - Research Site, Kōtoku
  - Research Site, Kyoto
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Nishinomiya-shi
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Ota-shi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shinagawa-ku
  - Research Site, Shinjuku-ku
  - Research Site, Tsukuba
  - Research Site, Yokohama
- Research Site, San Juan, Puerto Rico
- South Korea (5):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (8):
  - Research Site, Barcelona
  - Research Site, Bilbao (Vizcaya)
  - Research Site, Elche(Alicante)
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Palma de Mallorca
  - Research Site, Toledo
  - Research Site, Valencia
- Sweden (3):
  - Research Site, Stockholm
  - Research Site, Sundsvall
  - Research Site, Uppsala
- Taiwan (6):
  - Research Site, Hsinchu
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
  - Research Site, Yung Kang City
- United Kingdom (11):
  - Research Site, Cambridge
  - Research Site, Cardiff
  - Research Site, Edinburgh
  - Research Site, Greater London
  - Research Site, London
  - Research Site, Londonderry
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Portsmouth
  - Research Site, Surrey
  - Research Site, Taunton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Bardia A, Pusztai L, Albain K, Ciruelos EM, Im SA, Hershman D, Kalinsky K, Isaacs C, Loirat D, Testa L, Tokunaga E, Wu J, Dry H, Barlow W, Kozarski R, Maxwell M, Harbeck N, Sharma P. TROPION-Breast03: a randomized phase III global trial of datopotamab deruxtecan +/- durvalumab in patients with triple-negative breast cancer and residual invasive disease at surgical resection after neoadjuvant therapy. Ther Adv Med Oncol. 2024 Apr 29;16:17588359241248336. doi: 10.1177/17588359241248336. eCollection 2024. PMID 38686016
- See also: Breast Cancer Study Locator details (for US) — https://www.breastcancerstudylocator.com/trial/listing/369195